CLINICAL TRIAL: NCT03243214
Title: Effect of Excitatory Theta-Burst Transcranial Magnetic Stimulation on Cognition in Patients With Both Parkinson's Disease and Mild Cognitive Impairment and Analysis of Functional and Structural Brain Changes After Stimulation
Brief Title: Effect of Transcranial Magnetic Stimulation on Cognition and Neural Changes in Parkinson's Disease
Acronym: PD-MCI-TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Montreal Neurological Institute and Hospital (Other); McGill University (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Oury Monchi, Professor and Tourmaline Chair in Parkinson's Disease, University of Calgary
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: REB15-1689
Record Dates: First submitted 2017-08-02; First posted 2017-08-08 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Parkinson's Disease; Mild Cognitive Impairment
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a randomized double blind trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant and investigator do not know what treatment is applied (TMS stimulation or Sham-TMS stimulation with a different coil).
  The outcomes assessor will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-MCI, TMS (Active Comparator): The patient is treated with TMS stimulation according to protocol with an active coil.
  Interventions: Device: TMS
- PD-MCI, Sham-TMS (Sham Comparator): The patient is treated with Sham-TMS stimulation according to protocol with an inactive coil.
  Interventions: Device: Sham-TMS

INTERVENTIONS:
Device: TMS — Real or Sham TMS will be given to the PD-MCI patient
  Other Names: Magstim
  Arms: PD-MCI, TMS
Device: Sham-TMS — Real or Sham TMS will be given to the PD-MCI patient
  Arms: PD-MCI, Sham-TMS

SUMMARY:
Parkinson's disease (PD) affects more than 100,000 Canadians and results in symptoms affecting both motor and cognitive (thinking and memory) functions. Parkinson's disease with Mild Cognitive Impairment (MCI) frequently results in development of dementia for which few treatment options exist. Transcranial Magnetic Stimulation (TMS) is used to alter activity in the outer regions of the brain and has been shown in previous studies to increase cognitive performance in patients with different disorders. This study will investigate the effectiveness of TMS as a clinical treatment for the cognitive deficits associated with Parkinson's disease. 64 male and female participants between the ages of 50 and 90 will attend eight study visits over a period of 63 to 66 days. This study is a double-blind randomized clinical trial meaning the participant will be assigned by chance to either the TMS-treatment group or the Sham-treatment group. Additionally, a combination of memory and thinking tests and Magnetic Resonance Imaging (MRI) will be used to see if there are structural and functional changes within the brain. Genotyping and blood analysis before and after treatment for different biomarkers will also be performed and these data will be compared to the TMS data. Initially, this research will increase knowledge about the effects of TMS on various brain regions. Ultimately, we will be able to determine if TMS can be used as a complementary therapy for PD to improve cognitive performance and to reduce progression into dementia.

DETAILED DESCRIPTION:
Visit 1:

Informed Consent Neuropsychological Battery

Visit 2: (1-2 days later) Blood Draw Neuropsychiatric Assessment Questionnaires Companion Questionnaire to take home UPDRS

Visit 3: (up to a week after visit 2) MRI Scan while performing Executive Task

Visit 4: (1-3 days after visit 3) TMS- or Sham-Treatment (two sessions , 20 min each, 1 hour apart)

Visit 5: (2-3 days after visit 4) Same as Visit 4

Visit 6: (2-3 days after visit 5) Same as Visit 4

Visit 7: (1 day after visit 6) Neuropsychological Battery UPDRS

Visit 8: (1 day after visit 7) MRI Scan while performing Executive Task Blood Draw

Visit 9: (1 month after visit 6) Neuropsychological Battery UPDRS

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease any stage
* Mild Cognitive Behaviour confirmed through neuropsychological assessment
* MRI Compatibility

Exclusion Criteria:

* Alcohol-dependency
* Severe psychiatric disorder, neurological disorder, epilepsy or stroke
* General anaesthesia in the past six months
* History of cerebrovascular disorders
* Colour-blindness

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
TMS stimulation applied to the left DLPFC has a quantifiable effect on cognition | Neuropsychological Assessments: Baseline, one day after and one month after TMS stimulation
  Changes in one or more of the five assessed brain domains at baseline and one day after stimulation will be measured by comparing the scores for the different neuropsychological tests.
  The same neuropsychological assessment one month after TMS stimulation will show, if possible changes from one day after are longer lasting and can still be seen.

SECONDARY OUTCOMES:
Change in structural grey and white matter in the brain at baseline compared to after TMS stimulation | MRI: Baseline and two days after TMS stimulation
  MRI analysis will measure any changes in cortical thickness (mm) or other structural changes in the brain after TMS or Sham-TMS stimulation
Change in executive functioning measured as BOLD fMRI sequence | MRI: Baseline and two days after TMS stimulation
  The executive task, Wisconsin Card Sorting Task, will be performed in the scanner to measure the level of activation in the basal ganglia and the prefrontal cortex via BOLD functional MRI sequence to see changes after TMS stimulation compared to baseline.
Change in levels of biomarkers of interest (alpha-synuclein and BDNF) in serum after TMS stimulation compared to baseline. | Blood draws: Baseline and two days after TMS stimulation
  Measure the concentration of alpha-synuclein and BDNF in serum at baseline and after TMS stimulation with the Meso Scale Discovery method. These assays are highly developed ELISA assays using electrochemiluminescence.
Genotyping | Blood draw for DNA analysis: Baseline
  Analyze DNA for following genes: COMT, DAT1, MAPT, ApoE, GBA, CHCRA4, SNCA, BDNF These genes of interest will be correlated to changes in the neuropsychological assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Oury Monchi, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Department of Clinical Neurosciences, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Lang S, Gan LS, Yoon EJ, Hanganu A, Kibreab M, Cheetham J, Hammer T, Kathol I, Sarna J, Martino D, Monchi O. Theta-Burst Stimulation for Cognitive Enhancement in Parkinson's Disease With Mild Cognitive Impairment: A Randomized, Double-Blind, Sham-Controlled Trial. Front Neurol. 2020 Dec 21;11:584374. doi: 10.3389/fneur.2020.584374. eCollection 2020. PMID 33408684